CLINICAL TRIAL: NCT04720547
Title: Sleep and Breathing in Health and Disease (Part 2A - Chemical Stimuli, Sleep and Breathing in the General Population)
Brief Title: Sleep and Breathing in the General Population - Chemical Stimuli
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, M Safwan Badr, Chair of Internal Medicine, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1203010749; 5R01HL130552-05 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Results first posted 2022-04-28 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Sleep-disordered Breathing
Keywords: Sleep-disordered Breathing; central sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central | interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: After an initial assessment to determine eligibility, participant complete two in-lab night studies in a randomized manner including one night with the administration of zolpidem and another without zolpidem.
Who Masked: Outcomes Assessor
Masking Description: Personnel conducting assessment of outcomes and data analysis are blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zolpidem, then No Treatment (Experimental): Participants will be administered zolpidem for the first night study, and No Treatment during the second night study.
  Interventions: Drug: Zolpidem; Other: No Treatment
- No Treatment, then Zolpidem (Experimental): Participants will be administered zolpidem for the second night study, and No Treatment during the first night study.
  Interventions: Drug: Zolpidem; Other: No Treatment

INTERVENTIONS:
Drug: Zolpidem — A nonbenzodiazepine hypnotic
  Other Names: Ambien
Other: No Treatment — The Control condition in which participants do not receive medication.

SUMMARY:
Central sleep apnea (CSA) is a common condition and its treatment remains elusive. The focus of this proposal is to identify the role of the physiologic path involving cortical arousals in CSA by decreasing arousal frequency using the pharmacological agent zolpidem. The goal is to identify the acute effects of administering zolpidem on sleep and respiratory outcomes, and subsequently, its effect on the severity of CSA and propensity to develop CSA. This study will shed light on the mechanisms underlying CSA that involve cortical arousals and will guide future therapeutic interventions for CSA.

DETAILED DESCRIPTION:
The literature suggests that zolpidem may be effective in the treatment of central sleep apnea (CSA). However, evidence regarding the efficacy of zolpidem and the underlying mechanisms involved in its effect on CSA are not well-studied. Furthermore, respiratory-related arousals are hypothesized to contribute CSA symptoms and severity. The aim of the study is to determine the effect of decreasing respiratory-related arousals on the propensity to develop central apnea. The investigators hypothesize that administration of the nonbenzodiazepine hypnotic zolpidem will decrease the frequency of respiratory-related arousals, lower the central apnea-hypopnea index, and widen the CO2 reserve during sleep in patients with CSA compared to no treatment. Participants will complete a night study on a low dose of zolpidem and another night study without zolpidem in a crossover manner. The order of night studies is randomized. The results will help unveil the role of arousals in CSA and the acute effect of zolpidem on CSA severity and the propensity to CSA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women Veterans with central sleep apnea, defined as Apnea Hypopnea Index (AHI)>15/hour with CAHI>5/hour, will be included in the experiments.

Exclusion Criteria:

* less than 18 years old
* pregnant or breastfeeding female
* have severe respiratory disease that require to be on oxygen
* recent health event that may affect the ability to participate in the study,
* Body Mass Index (BMI) is >40 kg/m2
* significant insomnia
* mental instability
* recent health event that may affect sleep
* if at any time the principal investigator (PI) identifies that a certain drug is not suitable, or are unable to use the device that is used to treat sleep apnea, will be not be allowed to participate in the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Safwan Badr, MD, MBA, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmad B, Sankari A, Eshraghi M, Aldwaikat A, Yarandi H, Zeineddine S, Salloum A, Badr MS. Effect of Zolpidem on nocturnal arousals and susceptibility to central sleep apnea. Sleep Breath. 2023 Mar;27(1):173-180. doi: 10.1007/s11325-022-02593-3. Epub 2022 Mar 14. PMID 35286569

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Zolpidem, Then No Treatment: Participants will be administered zolpidem for the first night study, and No Treatment during the second night study.
  Zolpidem: A nonbenzodiazepine hypnotic
- Experimental: No Treatment, Then Zolpidem: Participants will be administered zolpidem for the second night study, and No Treatment during the first night study.
Period: Overall Study
Arm/Group | Experimental: Zolpidem, Then No Treatment | Experimental: No Treatment, Then Zolpidem
Started | 6 | 8
Completed | 6 | 5
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem, Then No Treatment | No Treatment, Then Zolpidem | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] — The year of birth was acquired from the participant's medical record and the participant's age at the start of the study was calculated and included in the baseline measure.
  years | 56.7 (12.7) | 70.4 (4.3) | 62.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — The sex of participants was acquired from their medical records and confirmed with them through a baseline questionnaire before the beginning of the study.
  Participants
    Female | 2 | 0 | 2
    Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The ethnicity of participants was acquired through a baseline questionnaire before the beginning of the study. Participants indicated whether they identified as Hispanic/Latino, or non-Hispanic/latino, and were given the option to leave it blank.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 6 | 5 | 11
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race of participants was acquired through a baseline questionnaire before the beginning of the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 4 | 7
    White | 3 | 1 | 4
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Veteran Status: Yes [Count of Participants; unit: Participants] — This variable indicates whether the participant is an Army Veteran. Veteran status was determined from the participant's medical record and verified with the participant through a baseline questionnaire at the beginning of the study.
  Participants | 5 | 5 | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] — The body mass index was measured through a baseline questionnaire or acquired from the medical records and verified with participants.
  kg/m^2 | 29.6 (5.6) | 32.2 (4.8) | 30.8 (5.3)
Neck Girth [Mean (Standard Deviation); unit: cm] — Neck girth was measured at baseline.
  cm | 38.9 (6.2) | 41.4 (3.5) | 40.0 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: The Central Apnea-hypopnea Index
Description: The number of central apneas and hypopneas per hour of sleep was obtained from polysomnography studies.
Time Frame: one night
Measure: Mean (Standard Error); unit: events per hour
Groups:
- Zolpidem: Outcomes from the Zolpidem night for participants in both sequences
- No Treatment: Outcomes from the No Treatment night for participants in both sequences
Arm/Group | Zolpidem | No Treatment
Number analyzed (Participants) | 10 | 10
events per hour | 14.1 (4.4) | 29.9 (7.6)

2. Primary Outcome: Respiratory Arousal Index
Description: A measure of the frequency of respiratory-related arousals during sleep
Time Frame: one night
Measure: Mean (Standard Error); unit: events per hour
Arm/Group | Zolpidem | No Treatment
Number analyzed (Participants) | 10 | 10
events per hour | 23.3 (4.4) | 39.7 (7.7)

3. Secondary Outcome: CO2 Reserve
Description: CO2 reserve is the requisite change to induce central apnea is referred to as the CO2 reserve, which can be positive or negative. CO2 reserve is defined as the difference between the eupneic end-tidal CO2 pressure and the end-tidal CO2 pressure induced by the ventilation protocol that is sufficient to trigger a central apnea as defined by the American Academy of Sleep Medicine.
Time Frame: one night
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Zolpidem | No Treatment
Number analyzed (Participants) | 8 | 8
mmHg | -0.63 (2.42) | -0.44 (4.17)

4. Secondary Outcome: Controller Gain
Description: Controller gain is a ventilatory response to changes in end-tidal PCO2. Controller gain was calculated by dividing the difference in minute ventilation between the post-mechanical ventilation induced by the ventilation protocol and steady-state respiration by the difference in the end-tidal CO2 pressure between the mechanical ventilation and steady-state respiration.
Time Frame: one night
Measure: Mean (Standard Error); unit: L/min*mmHg
Arm/Group | Zolpidem | No Treatment
Number analyzed (Participants) | 5 | 5
L/min*mmHg | 2.39 (1.10) | 3.95 (2.34)

5. Secondary Outcome: Stead-State Plant Gain (mmHg
Description: Plant gain is a blood gas response to a change in ventilation. This measure represents the effectiveness of the "plant" in eliminating CO2. Steady-state plant gain was calculated from the ratio of end-tidal CO2 to minute ventilation during stable respiration.
Time Frame: one night
Measure: Mean (Standard Error); unit: mmHg*L/min
Arm/Group | Zolpidem | No Treatment
Number analyzed (Participants) | 8 | 8
mmHg*L/min | 4.78 (0.79) | 5.27 (1.0)

6. Secondary Outcome: Respiratory Arousal Threshold
Description: The nadir pressure in the upper airway (supra-glottic pressure) prior to the occurrence of an arousal
Time Frame: one night
Measure: Mean (Standard Error); unit: cmH2O
Arm/Group | Zolpidem | No Treatment
Number analyzed (Participants) | 4 | 4
cmH2O | -8.72 (4.20) | -8.25 (5.63)

ADVERSE EVENTS:
Time Frame: Adverse effects were recorded for the 24 hours following the administration of the study medication
Arm/Group | Zolpidem | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT04720547/Prot_SAP_000.pdf